CLINICAL TRIAL: NCT05662332
Title: A Phase 3, Parallel-Design, Open-Label, Randomized Control Study to Evaluate the Efficacy and Safety of LY3209590 Administered Weekly Using a Fixed Dose Escalation Compared to Insulin Glargine in Insulin-Naïve Adults With Type 2 Diabetes
Brief Title: A Study of Insulin Efsitora Alfa (LY3209590) Compared to Glargine in Adult Participants With Type 2 Diabetes Who Are Starting Basal Insulin for the First Time (QWINT-1)
Acronym: QWINT-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18261; I8H-MC-BDCW (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-12-15; First posted 2022-12-22 (Actual); Results first posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes; T2D
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Masking Description: Sponsor will be blinded throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Insulin Efsitora Alfa (Experimental): Participants received Insulin Efsitora Alfa (insulin efsitora; 500 U/ml) administered subcutaneously (SC) once weekly (QW) for 52 weeks, with titration using fixed-doses 100 U, 150 U, 250 U, and 400 U.
  Interventions: Drug: Insulin Efsitora Alfa
- Insulin Glargine (Active Comparator): Participants received insulin glargine (100 U/ml) administered SC once daily (QD) for 52 weeks with titration by standard sliding-scale dose adjustments.
  Interventions: Drug: Insulin Glargine

INTERVENTIONS:
Drug: Insulin Efsitora Alfa — Administered SC
  Other Names: LY3209590 and Basal Insulin-FC
  Arms: Insulin Efsitora Alfa
Drug: Insulin Glargine — Administered SC
  Arms: Insulin Glargine

SUMMARY:
The main purpose of this study is to determine the efficacy and safety of insulin efsitora alfa (LY3209590) administered weekly using a fixed dose escalation compared to insulin glargine in adults with type 2 diabetes (T2D) who are starting basal insulin therapy for the first time.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of T2D according to the World Health Organization criteria.
* Have an HbA1c of 7.0% to 10.0%, inclusive, at screening.
* Are on a stable treatment of at least 1 antihyperglycemic medication, for at least 3 months prior to screening, and willing to continue the stable treatment for the duration of the study.
* Are insulin naive

Exceptions:

* short-term insulin treatment for a maximum of 14 days, prior to screening, and
* prior insulin treatment for gestational diabetes.

Exclusion Criteria:

* Have a diagnosis of type 1 diabetes (T1D), latent autoimmune diabetes, or specific type of diabetes other than T2D, for example, monogenic diabetes, diseases of the exocrine pancreas, or drug induced or chemical-induced diabetes.
* Have a history of >1 episode of ketoacidosis or hyperosmolar state or coma requiring hospitalization within 6 months prior to screening.
* Have had severe hypoglycemia episodes within 6 months prior to screening.
* Have known hemoglobinopathy, hemolytic anemia or sickle cell anemia, or any other traits of hemoglobin abnormalities known to interfere with the measurement of HbA1c.
* Have had New York Heart Association Class IV heart failure or any of these cardiovascular conditions within 3 months prior to screening
* acute myocardial infarction
* cerebrovascular accident (stroke), or
* coronary bypass surgery.
* Have had gastric bypass (bariatric) surgery, restrictive bariatric surgery, for example Lap-Band, or sleeve gastrectomy within 1 year prior to screening
* Have had significant weight gain or loss within 3 months prior to screening, for example, ≥5%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 795 (Actual)
Dates: Start 2023-01-14 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2024-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (70):
- United States (39):
  - Cahaba Research, Birmingham, Alabama
  - Syed Research Consultants Llc, Sheffield, Alabama
  - AMCR Institute, Escondido, California
  - Velocity Clinical Research, Gardena, Gardena, California
  - National Research Institute - Huntington Park, Huntington Park, California
  - National Research Institute - Wilshire, Los Angeles, California
  - Diabetes Associates Medical Group, Orange, California
  - Encompass Clinical Research, Spring Valley, California
  - Millennium Clinical Trials, Thousand Oaks, California
  - University Clinical Investigators, Inc., Tustin, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Clinical Research of West Florida, Inc. (Clearwater), Clearwater, Florida
  - Suncoast Research Group, Miami, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Center for Advanced Research & Education, Gainesville, Georgia
  - Pacific Diabetes & Endocrine Center, Honolulu, Hawaii
  - Central Illinois Diabetes and Clinical Research a Division of Prairie Education and Research Cooperative, Springfield, Illinois
  - American Health Network of Indiana, LLC - Franklin, Franklin, Indiana
  - American Health Network of Indiana, LLC - Muncie, Muncie, Indiana
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division, Troy, Michigan
  - Clinvest Research LLC, Springfield, Missouri
  - University Of Nebraska Medical Center, Omaha, Nebraska
  - Mid Hudson Medical Research, New Windsor, New York
  - Meridian Clinical Research, LLC, Vestal, New York
  - Intend Research, LLC, Norman, Oklahoma
  - Decpa, Llc, Feasterville-Trevose, Pennsylvania
  - Office 18, Pittsburgh, Pennsylvania
  - WR-Clinsearch, LLC, Chattanooga, Tennessee
  - Private Practice - Dr. Osvaldo A. Brusco, Corpus Christi, Texas
  - Dallas Diabetes Research Center, Dallas, Texas
  - Prime Revival Research Institute, Flower Mound, Texas
  - Endocrine Associates, Houston, Texas
  - Endocrine Ips, Pllc, Houston, Texas
  - North Hills Family Medicine/North Hills Medical Research, North Richland Hills, Texas
  - Texas Valley Clinical Research, Weslaco, Texas
  - Eastside Research Associates, Redmond, Washington
- Argentina (21):
  - Centro de Investigaciones Metabólicas (CINME), Ciudad Autónoma de Buenos Aire, Buenos Aires
  - Instituto de Investigaciones Clínicas Mar del Plata, Mar del Plata, Buenos Aires
  - DIM Clínica Privada, Ramos Mejía, Buenos Aires
  - Go Centro Medico San Nicolás, San Nicolás de los Arroyos, Buenos Aires
  - Asociación de Beneficencia Hospital Sirio Libanés, Buenos Aires, Buenos Air
  - Stat Research S.A., Buenos Aires, Ciudad Aut
  - Centro Médico Viamonte, Buenos Aires, Ciudad Aut
  - Glenny Corp, Buenos Aires, Ciudad Aut
  - CEMEDIAB, C.a.b.a., Ciudad Aut
  - Investigaciones Medicas Imoba Srl, Buenos Aires, Ciudad Autónoma de Buenos Aire
  - CIPREC, Buenos Aires, Ciudad Autónoma de Buenos Aire
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada, Ciudad Autonoma de Buenos Aire, Ciudad Autónoma de Buenos Aire
  - Centro Medico Privado San Vicente Diabetes, Córdoba, Córdoba Province
  - Instituto Médico Río Cuarto, Río Cuarto, Córdoba Province
  - CIPADI - Centro Integral de Prevencion y Atencion en Diabetes, Godoy Cruz, Mendoza Province
  - Instituto Médico Fundación Grupo Colaborativo Rosario Investigación y Prevención Medica, Rosario, Santa Fe Province
  - Clínica Mayo, San Miguel de Tucumán, Tucumán Province
  - Fundación Respirar, Buenos Aires
  - CENUDIAB, Ciudad Autónoma de Buenos Aire
  - Centro de Diagnóstico y Rehabilitación (CEDIR), Santa Fe
  - Sanatorio Norte, Santiago del Estero
- Mexico (8):
  - Instituto Jalisciense de Investigacion en Diabetes y Obesidad, Guadalajara, Jalisco
  - Diseno y Planeacion en Investigacion Medica, Guadalajara, Jalisco
  - RM Pharma Specialists, Mexico City, Mexico City
  - Instituto de Diabetes, Obesidad y Nutricion, Cuernavaca, Morelos
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León
  - Unidad Médica para la Salud Integral, San Nicolás de los Garza, Nuevo León
  - Medical Care and Research SA de CV, Mérida, Yucatán
  - Investigacion En Salud Y Metabolismo Sc, Chihuahua City
- Puerto Rico (2):
  - Ponce Medical School Foundation Inc., Ponce
  - Latin Clinical Trial Center, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the United States (US) and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Miller E, Davidson MB, Bajaj HS, Rosenstock J, Philis-Tsimikis A, Bergenstal RM, Case M, Ilag L, Threlkeld R, Levasseur E, Gelsey F. Evaluation of Overall Health State, Treatment Burden, and Satisfaction with Insulin Efsitora Alfa (Efsitora) vs. Daily Comparator in Adults with Type 2 Diabetes in the QWINT Clinical Trial Program. Diabetes Ther. 2026 Jan 27. doi: 10.1007/s13300-025-01833-5. Online ahead of print. PMID 41591636
- [Derived] Rosenstock J, Bailey T, Connery L, Miller E, Desouza C, Wang Q, Leohr J, Knights A, Carr MC, Child CJ; QWINT-1 trial investigators. Weekly Fixed-Dose Insulin Efsitora in Type 2 Diabetes without Previous Insulin Therapy. N Engl J Med. 2025 Jul 24;393(4):325-335. doi: 10.1056/NEJMoa2502796. Epub 2025 Jun 22. PMID 40548694
- See also: A Study of LY3209590 Compared to Glargine in Adult Participants With Type 2 Diabetes Who Are Starting Basal Insulin for the First Time (QWINT-1) — https://trials.lilly.com/en-US/trial/379581

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Insulin Efsitora Alfa | Insulin Glargine
Started | 397 | 398
Received at Least One Dose of the Study Drug | 397 | 398
Completed | 362 | 361
Not Completed | 35 | 37
Not completed — Death | 3 | 3
Not completed — Lost to Follow-up | 3 | 8
Not completed — Physician Decision | 1 | 2
Not completed — Protocol Deviation | 2 | 1
Not completed — Withdrawal by Subject | 14 | 14
Not completed — Assigned Treatment by Mistake | 5 | 7
Not completed — Non-compliance with study drug | 4 | 1
Not completed — Due to Bariatric surgery | 1 | 0
Not completed — Subject Moving out of State | 0 | 1
Not completed — Subject Missed the Schedule | 1 | 0
Not completed — The Patient Moved to Another City | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of the study drug.
Groups:
- Efsitora: Participants received Insulin Efsitora Alfa (insulin efsitora; 500 U/ml) administered subcutaneously (SC) once weekly (QW) for 52 weeks, with titration using fixed-doses 100 U, 150 U, 250 U, and 400 U.
- Glargine: Participants received Insulin glargine (100 U/ml) administered SC once daily (QD) for 52 weeks with titration by standard sliding-scale dose adjustments.
- Total: Total of all reporting groups
Arm/Group | Efsitora | Glargine | Total
Number analyzed (Participants) | 397 | 398 | 795
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.40 (10.02) | 56.20 (9.67) | 56.30 (9.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 194 | 203 | 397
  Male | 203 | 195 | 398
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 338 | 336 | 674
  Not Hispanic or Latino | 59 | 61 | 120
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 106 | 107 | 213
  Asian | 3 | 6 | 9
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 13 | 10 | 23
  White | 270 | 272 | 542
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Argentina | 170 | 171 | 341
  Mexico | 129 | 129 | 258
  United States | 98 | 98 | 196
HemoglobinA1c (HbA1c) [Mean (Standard Deviation); unit: Percentage of HbA1c] — HbA1c is the glycated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over the last 2-3 months. Population: All randomized participants who received at least one dose of the study drug and had HbA1c measurement at baseline.
  Percentage of HbA1c
    number analyzed (Participants) | 392 | 391 | 783
    (all) | 8.20 (0.91) | 8.28 (1.06) | 8.24 (0.99)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) [Noninferiority Analysis]
Description: HbA1c is the glycated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over the last 2-3 months. Least Squares (LS) Mean was determined using ANCOVA model with Baseline + Country + GLP-1 RA Use at Randomization Flag + Treatment (Type III sum of squares) as variables. Missing data at Week 52 were imputed by return-to-baseline multiple imputation approach.
Time Frame: Baseline, Week 52
Population: All randomized participants who received at least one dose of the study drug and had HbA1c measurement at baseline or Week 52, excluding participants discontinuing the study treatment due to inadvertent enrollment. All measurements were included regardless of the use of study treatment or rescue medication.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Efsitora | Glargine
Number analyzed (Participants) | 355 | 360
Percentage of HbA1c | -1.19 (0.0546) | -1.16 (0.0545)
Statistical Analysis 1: Comparison: Efsitora vs Glargine; Test type: Non-Inferiority — Noninferiority margin (NIM) was 0.4%; ANCOVA; LS Mean Change difference = -0.03, 95% CI 2-sided [-0.18 to 0.12]

2. Secondary Outcome: Change From Baseline in HbA1c [Superiority]
Description: HbA1c is the glycated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time. Least Squares (LS) Mean was determined using ANCOVA model with Baseline + Country + GLP-1 RA Use at Randomization Flag + Treatment (Type III sum of squares) as variables. Missing data at Week 52 were imputed by return-to-baseline multiple imputation approach.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Efsitora | Glargine
Number analyzed (Participants) | 355 | 360
Percentage of HbA1c | -1.19 (0.0546) | -1.16 (0.0545)
Statistical Analysis 1: Comparison: Efsitora vs Glargine; Test type: Superiority; p = 0.684, ANCOVA; LS Mean Change difference = -0.03, 95% CI 2-sided [-0.18 to 0.12]

3. Secondary Outcome: Change From Baseline in Fasting Glucose
Description: Change from baseline in fasting blood glucose measured by self-monitoring blood glucose (SMBG). LS mean was determined using ANCOVA model with Variable = Baseline + Country + GLP-1 RA Use at Baseline + Hemoglobin A1c Stratum at Baseline + Treatment (Type III sum of squares).
Time Frame: Baseline, Week 52
Population: All randomized participants who received at least one dose of the study drug and had a baseline and at least one post-baseline value for this outcome. Participants who discontinued the study drug due to inadvertent enrollment were excluded.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | Efsitora | Glargine
Number analyzed (Participants) | 341 | 359
milligrams per deciliter (mg/dL) | -46.76 (2.0797) | -50.92 (2.0595)
Statistical Analysis 1: Comparison: Efsitora vs Glargine; Week 52; Test type: Superiority; p = 0.155, ANCOVA; LS Mean Change difference = 4.16, 95% CI 2-sided [-1.58 to 9.90]

4. Secondary Outcome: Basal Insulin Dose at Week 52
Description: The insulin dose was recorded daily or weekly in an electronic diary. The average weekly basal insulin dose at Week 52 was reported. LS mean was determined using MMRM model with Baseline + Hemoglobin A1c Stratum at Baseline + Country + GLP-1 RA use at Randomization + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Week 52
Population: All randomized participants who received at least one dose of the study drug and had evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: Units per week (U/week)
Arm/Group | Efsitora | Glargine
Number analyzed (Participants) | 300 | 336
Units per week (U/week) | 289.1 (6.81) | 332.8 (6.68)
Statistical Analysis 1: Comparison: Efsitora vs Glargine; Week 52; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Change difference = -43.7, 95% CI 2-sided [-62.4 to -25.0]

5. Secondary Outcome: Rate Per Year of Hypoglycemia Events
Description: Rate of Composite Level 2 and 3 Hypoglycemia Events were reported. Hypoglycemia with glucose <54 mg/dL (Level 2) or Severe Hypoglycemia confirmed by the investigator to be an event that required assistance for treatment (Level 3) was reported. A severe hypoglycemic event is characterized by altered mental or physical status requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions for the treatment of hypoglycemia.
  Group mean was reported and determined by Negative binomial model using Number of episodes = Hemoglobin A1c at Baseline (%) + Treatment, with log (exposure in days/365.25) as an offset variable.
Time Frame: Baseline up to Week 52
Population: All randomized participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: Events per year
Arm/Group | Efsitora | Glargine
Number analyzed (Participants) | 397 | 398
Events per year | 0.50 (0.062) | 0.88 (0.152)
Statistical Analysis 1: Comparison: Efsitora vs Glargine; Test type: Superiority; p = 0.005, Negative binomial model; Relative Rate = 0.57, 95% CI 2-sided [0.39 to 0.84]

6. Secondary Outcome: Percentage of Participants With Hypoglycemia Events (Incidence)
Description: Incidence of hypoglycemic episodes is defined as 100 multiplied by the number of participants experiencing a hypoglycemic episode divided by the number of participants exposed to the study drug. Incidence of Composite Level 2 and 3 Hypoglycemia Events was reported. Hypoglycemic episodes are defined as an event that is associated with reported signs and symptoms of hypoglycemia with glucose <54 mg/dL (Level 2) or severe hypoglycemia confirmed by the investigator to be an event that required assistance for treatment (Level 3). A severe hypoglycemic event is characterized by altered mental or physical status requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions for the treatment of hypoglycemia.
Time Frame: Week 52
Population: All randomized participants who received at least one dose of the study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Efsitora | Glargine
Number analyzed (Participants) | 397 | 398
percentage of participants | 25.94 | 29.90

7. Secondary Outcome: Rate Per Year of Nocturnal Hypoglycemia Events
Description: The event rate of participant-reported clinically significant glucose <54 mg/dL (3.0 mmol/L) or severe nocturnal hypoglycemia that occurs at night and presumably during sleep between midnight and 6:00 AM), measured during treatment period up to week 52. Group mean is reported here. Group mean is determined by Negative Binomial Model using Number of episodes = .Hemoglobin A1c at Baseline (%) + Treatment, with log (exposure in days/365.25) as an offset variable.
Time Frame: Baseline up to Week 52
Population: All randomized participants who received at least one dose of the study drug.
Measure: Mean (Standard Error); unit: Events per year
Arm/Group | Efsitora | Glargine
Number analyzed (Participants) | 397 | 398
Events per year | 0.05 (0.013) | 0.08 (0.021)
Statistical Analysis 1: Comparison: Efsitora vs Glargine; Test type: Superiority; p = 0.155, Negative binomial model; Relative Rate = 0.58, 95% CI 2-sided [0.28 to 1.23]

8. Secondary Outcome: Percentage of Participants With Nocturnal Hypoglycemia Events (Incidence)
Description: Incidence of nocturnal hypoglycemic episodes is defined as 100 multiplied by the number of participants experiencing a hypoglycemic episode divided by the number of participants exposed to the study drug. Nocturnal hypoglycemia is defined as any hypoglycemic event that occurs between bedtime and waking. The event rate of participant-reported clinically significant glucose <54 mg/dL (3.0 mmol/L) or severe nocturnal hypoglycemia that occurs at night and presumably during sleep between midnight and 6:00 AM), measured during treatment period up to week 52..
Time Frame: Week 52
Population: All randomized participants who received at least one dose of the study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Efsitora | Glargine
Number analyzed (Participants) | 397 | 398
percentage of participants | 3.53 | 5.03

9. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from baseline in body weight was reported. LS mean was determined using ANCOVA model with Variable = Baseline + Country + GLP-1 RA Use at Baseline + Hemoglobin A1c Stratum at Baseline + Treatment (Type III sum of squares).
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Kilogram (kg)
Arm/Group | Efsitora | Glargine
Number analyzed (Participants) | 357 | 361
Kilogram (kg) | 3.86 (0.190) | 3.29 (0.189)
Statistical Analysis 1: Comparison: Efsitora vs Glargine; Test type: Superiority; p = 0.033, Mixed Models Analysis; LS Mean difference (Final Values) = 0.57, 95% CI 2-sided [0.047 to 1.10]

10. Secondary Outcome: Change From Baseline in Treatment-Related Impact Measure - Diabetes (TRIM-D) Total Score
Description: The TRIM-D is a self-administered instrument, which assesses the impact of diabetes treatment on participants' functioning and well-being across available diabetes treatments. The TRIM-D consists of 28 items, each assessed on a 5-point scale. The TRIM-D questionnaire consists of 5 sub-domains.
  Treatment Burden (6 items) Daily Life (5 items) Diabetes Management (5 items), Compliance (4 items), and Psychological Health (8 items), where each question is scored on a 1-5-point scale with a higher score indicating a better health state (less negative impact). Mean TRIM-D individual sub-domain scores and total scores are later transformed to a 0-100 scale for analysis. LS mean change in scores from baseline to 52 weeks for total score are presented here.
  LS mean was determined using MMRM model with BASELINE + Hemoglobin A1c Stratum at Baseline + Country + GLP-1 RA. Use at Randomization + Treatment + Time + Treatment*Time(Type III sum of squares) as variables.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Efsitora | Glargine
Number analyzed (Participants) | 341 | 342
Score on a scale | 15.4 (0.608) | 13.87 (0.607)
Statistical Analysis 1: Comparison: Efsitora vs Glargine; Week 52; Test type: Superiority; p = 0.071, Mixed Models Analysis; LS Mean difference (Final Values) = 1.56, 95% CI 2-sided [-0.13 to 3.25]

11. Secondary Outcome: Change From Baseline in Diabetes Treatment Satisfaction Questionnaire - Change Version (DTSQ-c)
Description: The DTSQ-c is a validated, patient-reported questionnaire designed to assess perceived changes in satisfaction with diabetes treatment over time. It is especially useful in clinical trials comparing a new treatment to a previous one. The DTSQ-c includes 8 items, each scored on a 7-point Likert scale ranging from -3 (Much less satisfied) to +3 (Much more satisfied). A score of 0 indicates no change in perception.
  This outcome reports three domains: (1) Perceived frequency of hypoglycaemia - lower scores reflect fewer perceived episodes; (2) Perceived frequency of hyperglycaemia - lower scores reflect fewer perceived episodes; (3) Treatment satisfaction -Aggregated score from the remaining 6 items assessing satisfaction with treatment, convenience, flexibility, understanding, and willingness to continue. A higher scores indicating greater improvement in satisfaction. Total score range: -18 to +18.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Efsitora | Glargine
Number analyzed (Participants) | 324 | 342
Score on a scale
  Perceived frequency of hypoglycemia score | -1.2 (1.95) | -1.3 (1.89)
  Perceived frequency of hyperglycemia score | -1.0 (1.84) | -0.9 (1.80)
  Treatment satisfaction score | 15.1 (4.57) | 14.5 (4.73)

12. Secondary Outcome: Percentage of Participants Reporting Treatment Experience Using the Simplicity of Diabetes Treatment Questionnaire (SIM-Q) Single Medication Status Version
Description: The SIM-Q is a brief 10-item measure developed to assess the simplicity and complexity of treatment for T2D. This version of the instrument assesses the simplicity and complexity of a single medication. Only the last 2 questions/items of the SIM-Q were completed by the study participants:
  1. "How simple or complex is your medication treatment for diabetes?"
  2. "Overall, how simple or complex is it to manage your diabetes, including medication, checking your blood glucose levels, diet, and any other aspects of diabetes treatment?" Participants were asked to provide responses to the study intervention at Week 52. Each item is scored on a 5-point scale ranging from "Very complex" to "Very simple." Higher scores indicate a more favorable (simpler) treatment experience.
Time Frame: Week 52
Population: All randomized participants who received at least one dose of the study drug and had evaluable data for this outcome. Participants who discontinued the study drug due to inadvertent enrollment were excluded.
Measure: Number; unit: Percentage of participants
Arm/Group | Insulin Efsitora Alfa | Insulin Glargine
Number analyzed (Participants) | 317 | 335
Percentage of participants
  SIMQF - How Simple or Complex Medication: Very Complex | 2.5 | 2.4
  SIMQF - How Simple or Complex Medication: Complex | 0.3 | 1.2
  SIMQF - How Simple or Complex Medication: A Little Complex | 6.0 | 6.6
  SIMQF - How Simple or Complex Medication: Simple | 37.2 | 41.2
  SIMQF - How Simple or Complex Medication: Very Simple | 53.9 | 48.7
  SIMQF - Overall How to Manage Diabetes: Very Complex | 1.6 | 3.0
  SIMQF - Overall How to Manage Diabetes: Complex | 4.7 | 4.8
  SIMQF - Overall How to Manage Diabetes : A Little Complex | 16.4 | 15.5
  SIMQF - Overall How to Manage Diabetes: Simple | 41.0 | 40.3
  SIMQF - Overall How to Manage Diabetes: Very Simple | 36.3 | 36.4

13. Secondary Outcome: Change From Baseline in Diabetes Injection Device Experience Questionnaire (DID-EQ) in Device Characteristics
Description: DID-EQ is a validated, self-administered, 10-item PRO instrument designed to assess participants' perceptions of diabetes injection delivery systems.This outcome measure reports only the Device Characteristics Subscale, which includes Items 1 through 7. These items evaluate specific features of injection devices such as:
  * Ease of preparation
  * Comfort during injection
  * Portability
  * Discreetness
  * Confidence in dose delivery
  * Ease of learning to use
  * Satisfaction with device features
  Each item is rated on a 4-point Likert scale: Strongly Disagree, Disagree, Agree, Strongly Agree. Responses are transformed to a 0-100 scale, where 0 represents most negative perception and 100 represents the most positive perception.Higher scores indicate more favorable perceptions of the injection device.
  LS Mean determined using ANCOVA model with Country + GLP-1 RA Use at Randomization + HbA1c Stratum at Baseline + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Efsitora | Glargine
Number analyzed (Participants) | 344 | 345
score on a scale | 91.4 (0.71) | 89.6 (0.71)
Statistical Analysis 1: Comparison: Efsitora vs Glargine; Week 52; Test type: Superiority; p = 0.072, Mixed Models Analysis; LS Mean difference (Final Values) = 1.8, 95% CI 2-sided [-0.2 to 3.8]

14. Secondary Outcome: Percentage of Participants in Treatment Experience in Diabetes Injection Device Experience Questionnaire (DID-EQ) (3-Global Items)
Description: The DID-EQ is a validated, self-administered, 10-item PRO instrument designed to assess participants' perceptions of diabetes injection delivery systems.
  This outcome measure specifically reports the summary of DID-EQ scores for the 3 global items:
  * Item 8: Overall satisfaction with the injection device
  * Item 9: Ease of use of the injection device
  * Item 10: Convenience of the injection device
  Each item is rated on a 4-point Likert scale:
  * Strongly Disagree
  * Disagree
  * Agree
  * Strongly Agree
  Responses are transformed to a 0-100 scale, where:
  * 0 = Most negative perception
  * 100 = Most positive perception
  Higher scores indicate more favorable perceptions of the injection device's global characteristics.
Time Frame: Week 52
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | Efsitora | Glargine
Number analyzed (Participants) | 344 | 345
percentage of participants
  Satisfied with the Injection Device (Strongly disagree) | 0.3 | 1.2
  Satisfied with the Injection Device (Disagree) | 0 | 0.3
  Satisfied with the Injection Device (Agree) | 15.4 | 19.1
  Satisfied with the Injection Device (Strongly Agree) | 84.3 | 79.4
  Easy to Use the Injection Device (Strongly disagree) | 0.3 | 0.9
  Easy to Use the Injection Device (Disagree) | 0 | 0.3
  Easy to Use the Injection Device (Agree) | 14.0 | 17.1
  Easy to Use the Injection Device (Strongly Agree) | 85.8 | 81.7
  Convenient to Use the Injection Device (Strongly disagree) | 0.3 | 1.2
  Convenient to Use the Injection Device (Disagree) | 0 | 0.3
  Convenient to Use the Injection Device (Agree) | 17.4 | 20.3
  Convenient to Use the Injection Device (Strongly agree) | 82.3 | 78.3

ADVERSE EVENTS:
Time Frame: Baseline up to Week 57
Description: All randomized participants who received atleast one dose of study drug. Participants were analyzed according to the treatment they were assigned. Gender specific events occurring only in male or female participants have had the number of participants at risk adjusted accordingly.
Arm/Group | Efsitora | Glargine
All-Cause Mortality (participants affected / at risk) | 3/397 | 3/398
Serious Adverse Events (participants affected / at risk) | 26/397 | 21/398
Other Adverse Events (participants affected / at risk) | 104/397 | 121/398
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Efsitora (N=397) | Glargine (N=398)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 2 (2)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 2 (2) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 2 (2)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Dermatofibrosarcoma protuberans (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebellar haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 1/194 (1) | 0/203 (0)
Adnexa uteri mass (Reproductive system and breast disorders) | 1/194 (1) | 0/203 (0)
Breast hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Prostatectomy (Surgical and medical procedures) | 0/203 (0) | 1/195 (1)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Efsitora (N=397) | Glargine (N=398)
Covid-19 (Infections and infestations) | 21 (21) | 9 (9)
Influenza (Infections and infestations) | 29 (30) | 23 (26)
Urinary tract infection (Infections and infestations) | 18 (20) | 25 (27)
Drug titration error (Injury, poisoning and procedural complications) | 13 (14) | 39 (53)
Headache (Nervous system disorders) | 20 (24) | 20 (24)
Hypertension (Vascular disorders) | 21 (24) | 16 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-05-31): https://cdn.clinicaltrials.gov/large-docs/32/NCT05662332/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-26): https://cdn.clinicaltrials.gov/large-docs/32/NCT05662332/SAP_001.pdf